CLINICAL TRIAL: NCT00000943
Title: A Controlled, Pilot Study of the Immunogenicity of Remune in HIV-Infected Subjects Receiving Either Highly Active Antiretroviral Therapy (HAART) Alone or HAART and Interleukin-2 (IL-2): A Nested Substudy of ACTG 328
Brief Title: A Study to Test If Giving Remune (an HIV Vaccine) Can Improve the Immune Systems of HIV-Positive Patients Who Are Also Participating in ACTG 328
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5046s; ACTG 328 (Main Study); AACTG A5046s; 10794 (Registry Identifier: DAIDS ES Registry Number); ACTG A5046s
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Lymphocytes; Interleukin-2; Drug Therapy, Combination; AIDS Vaccines; CD4 Lymphocyte Count; Cell Division; HIV Core Protein p24; Anti-HIV Agents; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Tetanus Toxoid; Hepatitis A Vaccines; HIV-1 immunogen, incomplete Freund's adjuvant; Hepatitis B Vaccines

INTERVENTIONS:
Biological: Tetanus Toxoid Vaccine
Biological: Hepatitis A Vaccine (Inactivated)
Biological: HIV-1 Immunogen
Biological: Hepatitis B Vaccine (Recombinant)

SUMMARY:
The purpose of this study is to determine the effects of an HIV vaccine (Remune) on the immune system. This study involves patients who have received at least 60 weeks of anti-HIV therapy, either alone or in combination with IL-2, while enrolled in ACTG 328.

Remune is an experimental HIV vaccine. To see how the body's immune system reacts, this vaccine will be given with 1 to 3 other vaccines, and skin tests will monitor the body's reaction.

DETAILED DESCRIPTION:
Proliferative responses to HIV antigens are either absent or of small magnitude in HIV-infected patients, even in the early stages of infection when vigorous proliferative responses to recall antigens are still seen. Remune consists of an inactivated, gp120-depleted virus intended to stimulate HIV-specific immune responses. Remune has been reported to increase lymphocyte proliferative responses to HIV antigens in patients with high CD4 cell counts. Many other T-cell-dependent responses are also impaired in HIV-infected patients, such as after vaccination with hepatitis A or B vaccine. In this study, patients with moderately advanced HIV disease who have already received 52 weeks of either HAART or HAART plus IL-2 are vaccinated with Remune and a control recall immunogen, tetanus toxoid (TT), to evaluate whether these patients can develop new CD4 T-cell and CD8 T-cell responses to HIV-related antigens. The antibody response to hepatitis A and hepatitis B vaccinations also will be explored.

Fifty patients are enrolled in this substudy; 17 from the HAART only arm (Arm I of ACTG 328) and 33 from the HAART plus either CIV or subcutaneous IL-2 arms (Arms II and III of ACTG 328). All patients are vaccinated 3 times with Remune and twice with TT. If patients are hepatitis A total antibody negative, they receive hepatitis A vaccine twice. Additionally, if patients are hepatitis B surface antigen negative, hepatitis B core antibody and surface antibody negative, they receive hepatitis B vaccine 3 times. Patients who are negative for all hepatitis markers receive hepatitis A and B vaccines.

Week 0 of A5046s begins at or after Week 64 of ACTG 328 (for patients in the HAART-only arm) or 4 weeks after the initiation of the seventh or any subsequent IL-2 cycle of ACTG 328 (for patients in any of the IL-2-containing arms). [AS PER AMENDMENT 9/16/99: Patients can be screened through Week 124 of ACTG 328.] Patients receive Remune at Weeks 0, 8, and 16 and TT at Weeks 0 and 8. Hepatitis A and/or B vaccines are also given at these times, if indicated. Blood and skin tests are performed at Weeks 0, 8, 16, and 24 to measure immune response and lymphocyte proliferative responses.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have completed at least 60 weeks of treatment on ACTG 328.
* Are willing to continue on their assigned ACTG 328 treatment until after they have completed 24 weeks on this substudy.
* Have a viral load less than or equal to 2,000 copies/ml.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an active opportunistic (HIV-related) infection.
* Are pregnant or breast-feeding.
* Have taken or are taking certain medications that are prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hernan Valdez, Study Chair; Michael Lederman, Study Chair
Locations (2):
- United States (2):
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Valdez H, Mitsuyasu R, Landay A, Sevin AD, Chan ES, Spritzler J, Kalams SA, Pollard RB, Fahey J, Fox L, Namkung A, Estep S, Moss R, Sahner D, Lederman MM. Interleukin-2 Increases CD4+ lymphocyte numbers but does not enhance responses to immunization: results of A5046s. J Infect Dis. 2003 Jan 15;187(2):320-5. doi: 10.1086/346056. Epub 2003 Jan 6. PMID 12552459